CLINICAL TRIAL: NCT03103516
Title: Epidural Decompression Surgery Within 24 Hours After Acute Spinal Cord Injury Improves Spinal Nerve Function: a Prospective, Multicenter, Non-randomized, Controlled Trial
Brief Title: Epidural Decompression Surgery Within 24 Hours After Acute Spinal Cord Injury Improves Spinal Nerve Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Baoguo Jiang, Principal Investigator, Peking University People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PekingUPH_003
Record Dates: First submitted 2017-04-01; First posted 2017-04-06 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: 200 acute spinal cord injury patients (complete and incomplete) will undergo pre-hospital treatment in the Beijing Emergency Medical Center and Beijing Red Cross Emergency Rescue Center, and will receive in-hospital treatment in the Peking University People's Hospital, Peking University Third Hospital, Beijing Friendship Hospital Affiliated to Capital Medical University, Chaoyang Hospital Affiliated to Capital Medical University, and Chinese PLA General Hospital, China. There were 100 patients undergoing epidural decompression surgery within 24 hours and 100 patients receiving surgery after 24 hours.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early epidural decompression group (Experimental): The patients will be assigned to early (within 24 hours after spinal cord injury) epidural decompression group (n=100) according to the patient's condition and operation time.
  Interventions: Procedure: early epidural decompression group
- delayed epidural decompression group (Experimental): The patients will be assigned to delayed (exceed 24 hours after spinal cord injury) epidural decompression group (n=100) according to the patient's condition and operation time.
  Interventions: Procedure: delayed epidural decompression group

INTERVENTIONS:
Procedure: early epidural decompression group — The patients will be assigned to early (within 24 hours after spinal cord injury) epidural decompression group (n=100) according to the patient's condition and operation time.
  Arms: early epidural decompression group
Procedure: delayed epidural decompression group — The patients will be assigned to delayed (exceed 24 hours after spinal cord injury) epidural decompression group (n=100) according to the patient's condition and operation time.
  Arms: delayed epidural decompression group

SUMMARY:
To compare the effects of early (within 24 hours) and delayed (exceed 24 hours) epidural decompression surgery on the recovery of spinal nerve function in patients with acute spinal cord injury (complete and incomplete) at postoperative 6 months.

DETAILED DESCRIPTION:
Whether early epidural decompression surgery can restore neurological function in patients with acute spinal cord injury (complete and incomplete), and an effective time window for epidural decompression, are still controversial.

This trial will verify whether early epidural decompression surgery is more conducive to the recovery of spinal nerve function in patients with acute spinal cord injury (complete and incomplete) compared with delayed surgery. This trial will begin in August 2017. Data analysis of 200 patients will be finished in December 2019. All results will be completed in December 2020. This trial will provide clinical evidences for the selection of timing of epidural decompression surgery in patients with complete and incomplete spinal cord injury.

Adverse events Adverse events will be obtained from patients or their legal representatives. Major adverse events will include: limb paralysis deterioration, re-operation, respirator use (more than 1 week), tracheostomy, septicemia, pneumonia, acute respiratory distress syndrome, atelectasis, other respiratory complications, wound infection (superficial and deep), urinary tract infection, other infections, gastrointestinal bleeding, peptic ulcer, intestinal obstruction, acute myocardial infarction, other heart events, pulmonary embolism, cerebrovascular complication, hepatic failure, renal failure, delirium and depression.

Statistical methods

1. All data will be analyzed using SPSS 19.0 software.
2. Normally distributed measurement data will be expressed as mean, SD, minimums, and maximums. Non-normally distributed measurement data will be expressed as the lower quartile (q1) and median and upper quartiles (q3). Count data will be presented as the percentage.
3. Measurement data among groups will be compared using two-sample t-test or Mann-Whitney U test.
4. Count data will be analyzed using chi square test or Fisher's exact test. Ranked data will be analyzed using Wilcoxon signed-rank test.

Sample size ASIA motor score is one of the main outcome measures. In accordance with a previous study (Chikuda et al., 2013), taking power = 0.8 with a significance level of α = 0.05, we will need 45 patients per group when the difference to be detected in the ASIA motor score between the groups is 12 points and the common standard deviation is 20. If we assume a patient loss rate of 20%, we will require 54 patients per group, totally 108 patients. We therefore aim to include 200 patients in accordance with previous conditions on acute spinal cord injury (complete and incomplete) treatment in participating units.

Data management

1. All data will be input into the spinal cord injury treatment database. After the completion of the study, the research group and third-party statistical staffs will carry out data collation and analysis.
2. The participating units are responsible for filling in the information database. Data consistency and logic will be checked by computer program combined with manual review. Any questions will be answered by the person in charge of the project and the main staff, and returned to the data management center, and then the data manager will modify and update the database.
3. All inspection procedures need to be repeated several times until there is no doubt. All changes and updates are required for recording and filing. It is strictly forbidden to use correction fluid or correction tape. All researchers are required to ensure that the data recorded in the case report forms are authentic.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury patients will be evaluated as complete or incomplete (contusion) after admission using rectal examination, in accordance with American Spinal Injury Association and International Medical Society of Paraplegia (2000);
* Final diagnosis by spine CT and/or MRI;
* Cervical, thoracic and thoracolumbar fracture dislocation or without fracture dislocation but combined with spinal cord injury;
* No other injury involving life, injury severity score < 16;
* No anesthesia contraindication;
* No local skin infection, no severe soft tissue contusion, soft tissue condition of the operation area met the operation requirements;
* Age: 16-85 years old, irrespective of sex.

Exclusion Criteria:

* Active or recent severe infection
* Severe infectious diseases that need to be treated in infectious disease hospital;
* History of mental illness;
* History of metal allergy;
* Long-term alcohol abuse and drug abuse;
* Do not agree to participate in this trial; the legal representative of the patient refuses to sign informed consent;
* Poor compliance, cannot be followed up as required.

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
American Spinal Injury Association (ASIA) motor and sensory scores | at postoperative 6 months
  To assess spinal nerve function. Evaluation criteria for neurological function after spinal cord injury: Neurological function will be evaluated in accordance with American Spinal Injury Association and International Medical Society of Paraplegia (2000).

SECONDARY OUTCOMES:
American Spinal Injury Association (ASIA) impairment scale | changes of week 1, month 1 and month 3 after surgery
  to assess spinal nerve function
Evaluation of the incidence of complications | changes of week 1, month 1, month 3 and month 6 after surgery
  to assess the incidence of complications.The percentage of the number of cases of postoperative complications to total cases will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Baoguo Jiang, Ph.D, Principal Investigator — Department of Orthopedics, Peking University People's Hospital, Beijing, China
Locations (4):
- China (4):
  - Chaoyang Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital Affiliated to the Capital University of Medical Sciences, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sizheng Z, Boxuan H, Feng X, Dianying Z. A functional outcome prediction model of acute traumatic spinal cord injury based on extreme gradient boost. J Orthop Surg Res. 2022 Oct 12;17(1):451. doi: 10.1186/s13018-022-03343-7. PMID 36224595